CLINICAL TRIAL: NCT04070209
Title: The Role of Therapeutic Layering of Stereotactic Body Radiotherapy on Darolutamide in the Management of Oligoprogressive Castration Resistant Prostate Cancer: a Pilot Phase II Trial
Brief Title: Management of Oligoprogressive Castration Resistant Prostate Cancer (PCS X)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tamim Niazi, Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCS X
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Prostate Cancer; Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Darolutamide (BAY1841788)+ SBRT (Experimental): CRPC subjects will receive LHRH agonist in combination with the new generation of hormonal therapy Darolutamide (300mg).
  Subjects who progress on LHRH + Darolutamide and develop oligometastases will receive SBRT
  Interventions: Drug: Darolutamide (BAY1841788); Radiation: SBRT

INTERVENTIONS:
Drug: Darolutamide (BAY1841788) — Darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equivalent to a total daily dose of 1200 mg.
  Other Names: ODM-201
Radiation: SBRT — SBRT will consist of 2-5 fractions of highly targeted radiation therapy delivered every other day. The radiation component will be completed in 4-10 days.

SUMMARY:
This is the first pilot phase II trial assessing the response of SBRT layered on Darolutamide (BAY1841788) on RPFS and deferring palliative second line systemic therapy in M0CRPC with oligoprogression.

DETAILED DESCRIPTION:
Metastases-directed therapy with stereotactic body radiation therapy (SBRT) is emerging as a new treatment option for solid tumor patients with a limited number of metastases (< 5) at the time of recurrence/progression, so called oligoprogression therapy. As such, oligoprogression is defined as prostate cancer patients with castration resistance and no metastases (M0CRPC) who are receiving ADT and new generation hormonal therapy (enzalutamide, apalutamide or darolutamide) as standard of care, and who are then progressing to oligometastases. The new generation hormonal therapy used in this study will be darolutamide (ODM-201). The rationale behind this approach has been to delay the start of palliative systemic therapies that are most often toxic and associated with a negative impact on patient's quality of life, as well as being more costly. However, to date, there are no prospective published data or ongoing studies that are looking into non metastatic castration resistant prostate cancer (M0CRPC) patients who progress to oligometastases (oligoprogression). To this end, we are proposing this pilot phase II trial to assess the impact of SBRT on radiological progression-free survival (RPFS) of M0CRPC patients who are receiving darolutamide and progress to oligometastatic disease (oligoprogression).

Prostate cancer patients with castration resistance and no metastases (M0CRPC) diagnosed by bone scan and CT scan or MRI will be recruited in this phase II and initiate darolutamide while continuing on ADT (Part 1 of the study), if not receiving darolutamide prior to study entry already. Patients who then progress to wide spread metastases or metastases situated at locations not amenable to ablative therapy will be excluded and treated with second line therapy as per the treating physician. Patients with oligoprogression (< 5 mets) and amenable to ablative therapy will be then treated with SBRT or surgery as an ablative therapy if SBRT is not feasible (Part 2 of the study). All patients will continue to receive non-interrupted LHRH agonist, PSA testing every 6-12 weeks and re-imaging every 6 months. Imaging will also be repeated at the appearance of symptoms or at PSA progression, whichever occurs first and this schedule continues until disease progression.

This is the first pilot phase II trial assessing the response of SBRT layered on darolutamide on RPFS and deferring palliative second line systemic therapy in M0CRPC with oligoprogression. This phase II will consist of 66 M0CRPC patients treated with darolutamide, of which we anticipate 48 will be eligible for SBRT.

ELIGIBILITY:
Inclusion Criteria (Part 1):

* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features;
* M0CRPC at study entry defined as follows:

  1. Ongoing androgen deprivation therapy with a LHRH agonist or bilateral orchiectomy (i.e., surgical or medical castration);
  2. Serum testosterone level ≤ 1.7 nmol/L (50 ng/dL) at the Screening visit;
  3. PSA progression defined by a minimum of two subsequent rising PSA levels with an interval of ≥ 1 week between each determination. Patients who received an anti-androgen must have progression after withdrawal (≥ 4 weeks since last flutamide or ≥ 6 weeks since last bicalutamide or nilutamide). The PSA value at the Screening visit should be ≥ 2 μg/L (2 ng/mL)
  4. PSA doubling time of 10 months or less,
  5. M0 assessed by conventional imaging (CT/MRI + bone scan).

NOTE: If darolutamide started prior to study entry, evidence of inclusion criteria 1-5 listed above prior to start of darolutamide must be submitted to determine study eligibility

* Prior cytotoxic chemotherapy for prostate cancer in adjuvant setting post radical therapy is allowed;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 or Karnofsky performance status of > 80% or higher;
* Estimated life expectancy of ≥ 6 months;
* Ability to swallow the study drug whole and comply with study.
* Patients should not have been previously exposed to other ARATs (Abiraterone, Enzalutamide, Apalutamide)

Inclusion Criteria (Part 2):

* ≤ 5 metastatic sites (on conventional imaging);
* ≤ 4 tumors within any given organ system, excluding brain (e.g. up to 4 bone metastases, or 4 lung metastases);
* All sites of disease must be amenable to SBRT with no history of the metastases being irradiated (radiation exposure prior to the development of the metastases is permitted as long as the radiation exposure was not intended for the metastases. For example, if there is prior pelvic radiation to the prostate and a subsequent iliac metastasis develops within the previously irradiated pelvic radiation field, then the iliac metastasis would be eligible per the institution policy and practice);
* In the case of a suspicious lesion in an unusual location such as lung or thoracic lymph nodes (without other abdominal lymph nodes), a confirmatory imaging or biopsy is strongly recommended;

Exclusion Criteria (Part 1):

* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment;
* Presence of distant metastasis, including previously treated (clinical stage M1) is exclusive, however isolated pelvic nodal disease below the iliac bifurcation (clinical stage N1) is not an exclusion criteria.
* History of another malignancy within the previous 5 years other than curatively treated non-melanoma skin cancer;
* Absolute neutrophil count < 1,500/μL, platelet count < 100,000/μL, or hemoglobin < 5.6 mmol/L (9 g/dL) at the Screening visit (NOTE: patients may not have received any growth factors within 7 days or blood transfusions within 28 days of the hematologic laboratory values obtained at the Screening visit);
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal and total bilirubin > 1.5 times the upper limit of normal at the Screening visit;
* Creatinine > 2 times the upper limit of normal at the Screening visit;
* Clinically significant cardiovascular disease including:

  1. Stroke or myocardial infarction within 6 months;
  2. Uncontrolled angina within 6 months;
  3. Coronary/peripheral artery bypass graft within 6 months;
  4. Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patients with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan performed within three months results in a left ventricular ejection fraction that is ≥ 45%;
  5. History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
  6. Uncontrolled hypertension as indicated by a resting systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg at screening. Patients may be re-screened after adjustments of antihypertensive medications;
  7. Bradycardia as indicated by a heart rate of < 50 beats per minute on the Screening ECG;
* Gastrointestinal disorder or procedure which expects to interfere significantly with absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months);
* Major surgery within 4 weeks of enrollment (Day 1 Visit);
* Active viral hepatitis, active human immunodeficiency virus (HIV) or chronic liver disease
* Use of opiate analgesics (eg. morphine, fentanyl, etc.) for pain from prostate cancer within 4 weeks of enrollment (Day 1 visit). This does not apply to non-morphine drugs like codeine;
* Radiation therapy for treatment of the primary tumor within 3 weeks of enrollment (Day 1 visit);
* Radiation or radionuclide therapy for treatment of metastasis;
* Primary disease not treated;
* Hormone naïve prostate cancer patients;
* Treatment with estrogens or AR inhibitors (bicalutamide, flutamide, nilutamide, cyproterone acetate) within 4 weeks of enrollment (Day 1 visit);
* Treatment with systemic biologic therapy for prostate cancer (other than approved bone targeted agents and GnRH-analogue therapy) or other agents with anti-tumour activity within 4 weeks of enrollment (Day 1 visit);
* Prior use of an investigational agent that blocks androgen synthesis (e.g., abiraterone acetate, enzalutamide, Apalutamide, TAK-700, TAK-683, TAK-448) or targets the androgen receptor (e.g., BMS 641988) on clinical trials;
* Known or suspected contraindications or hypersensitivity to darolutamide or GnRH agonists or any of the components of the formulations;
* Use of an investigational agent within 4 weeks of enrollment (Day 1 visit);
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within four weeks of enrollment (Day 1 visit);
* Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data;
* Unable to swallow study medications and comply with study requirements

Exclusion criteria (Part 2):

* Known or suspected brain metastasis or active leptomeningeal disease;
* > 5 metastasis;
* More than 4 metastasis in the same organ;
* Patients considered for SBRT in previous history of radiation therapy to the same area.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-free Survival | 5 years
  Time from first day of SBRT until confirmed second radiological progression or start of new antineoplastic therapy

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy-Prostate | 5 years
  Evaluate the impact of the treatment on the patient's quality of life using the FACT-P questionnaire
Quality of Life - Fatigue | 5 years
  Evaluate the impact of the treatment on the patient's quality of life using the Brief Fatigue Inventory (BFI) questionnaire
Quality of Life - Pain | 5 years
  Evaluate the impact of the treatment on the patient's quality of life using the Brief Pain Inventory (BPI) questionnaire
Toxicity of ODM-201 | 5 years
  To determine acute and late toxicity due to ODM-201, scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time to Subsequent Systemic Antineoplastic Therapy | 5 years
  Time to the administration of subsequent antineoplastic systemic therapy
PSA response | 5 years
  PSA value and onset of biochemical failure will be recorded
Overall Survival | 5 years
  Time from randomization until death from any cause
Disease Specific Survival | 5 years
  Time from randomization until death due to prostate cancer
Time to Skeletal-related Event (SRE) | 5 years
  Date of first SRE will be recorded
Local Control | 5 years
  To evaluate the impact of SBRT on oligometastases progression by radiographic imaging or the start of new antineoplastic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Niazi, MD, Principal Investigator — Jewish General Hospital
Locations (10):
- Canada (10):
  - Prostate Cancer Centre, Calgary, Alberta
  - Centre of Applied Urology Research, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Service d'urologie et Centre de la prostate, Longueuil, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Sir Mortimer JGH, Montreal, Quebec
  - L'Hôtel-Dieu de Québec (CHUQ), Québec, Quebec
  - Hôpital Fleurimont (CHUS), Sherbrooke, Quebec
  - Centre hospitalier affilié universitaire régional (CHAUR), Trois-Rivières, Quebec